CLINICAL TRIAL: NCT03518138
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Q-122 for the Treatment of Vasomotor Symptoms in Female Breast Cancer Patients/Survivors Taking Tamoxifen or an Aromatase Inhibitor
Brief Title: Safety/Efficacy of Q-122 in Breast Cancer Patients Taking Tamoxifen or Aromatase Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Que Oncology (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q122-2001
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Vasomotor Symptoms (VMS)
MeSH Terms: interventions — N,N'-(1,4-phenylenebis(methylene))dipyrimidin-2-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1, study drug (Experimental): 65 patients treated with Q-122, 100 mg BID
  Interventions: Drug: Q-122
- Group 2, placebo (Placebo Comparator): 65 patients treated with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Q-122 — oral capsule of Q-122
  Arms: Group 1, study drug
Drug: Placebo — oral capsule of placebo
  Arms: Group 2, placebo

SUMMARY:
This is a Phase 2 proof-of-concept (POC) study designed to determine the effectiveness of Q-122 for the treatment of Vasomotor Symptoms (VMS) versus placebo. Participants who meet all eligibility criteria following the Screening/Run-In period will be randomized to 1 of 2 treatment arms; blinded Q-122 or placebo for a period of 28 days. All participants will be followed for a 2-week, drug-free, follow-up period after their last dose of blinded Q-122/placebo before termination from the study.

DETAILED DESCRIPTION:
Vasomotor symptoms (VMS) are significant in postmenopausal women with the most effective medications for relief being hormonal preparations. Non-hormonal medications have demonstrated efficacy but at a far lower level than estrogen replacement therapy. For women with a history of breast cancer, hormone replacement therapy is often contraindicated and is not an option for women receiving endocrine therapy including tamoxifen (TAM) and aromatase inhibitors (AI). Breast cancer survivors, and women receiving endocrine therapy in particular, have a high rate of problematic hot flashes. In an open label Phase 1 study of the safety and activity of Q-122 in breast cancer patients taking TAM or an AI, 8 of 9 women who received at least 1 dose of 100 mg and 10 of 11 women who received at least 1 dose of 200 mg had a reduction in hot flashes of 2 or more per day, the FDA criteria for anti-VMS activity. This study will define the effect of Q-122 versus placebo in a population of women with a history of or current breast cancer who have an average of 50 or more moderate to severe hot flashes per week.

ELIGIBILITY:
Inclusion Criteria:

1. Be a female, aged between 18 - 70 years on the day of informed consent.
2. Have a history of or current breast cancer and currently taking tamoxifen or an aromatase inhibitor.
3. On a stable dose of TAM or an AI for a minimum of 30 days before the Screening Visit and no anticipated need to change the dose for the duration of the study.
4. Experience an average of at least 50 moderate to severe hot flashes/week for the 2 weeks immediately preceding the Run-In Visit (i.e., during the Screening period).
5. If on thyroid medication, on a stable dose for a minimum of 30 days before the Screening Visit and no anticipated need to change the dose for the duration of the study.
6. Willing and able to complete the daily participant diary, attend all study visits, and participate in all study procedures.
7. Able to provide informed consent.

Exclusion Criteria:

1. Childbearing potential, pregnancy, or lactation except in patients who are on stable dose of AI in combination with luteinizing hormone releasing hormone agonists such as Zoladex, Leuprolide (Lupron) or equivalent. Non-childbearing potential is defined as physiologically incapable of becoming pregnant by one of the following:

   * Has had a partial or complete hysterectomy or
   * Has had a bilateral oophorectomy or
   * Has had a bilateral tubal ligation or fallopian tube inserts or
   * Is post-menopausal (amenorrhea > 1 year) confirmed by levels of follicle stimulating hormone (FSH). FSH levels may be lower in menopausal women treated with tamoxifen when compared with FSH levels appropriate for confirming menopause in women not treated with tamoxifen. For those patients who are on stable dose of tamoxifen, confirmation of menopause is based on the clinical opinion of the PI and medical monitor on a 'case-by-case basis'.
2. Currently experiencing undiagnosed vaginal bleeding.
3. Women with advanced breast cancer (Stage 4).
4. Greater than 60% reduction in the frequency of moderate to severe hot flashes during the 1-week single blind Run-In period or inability to correctly record hot flashes and/or drug dosing in the participant diary.
5. Participation in another clinical or surgical trial within 30 days prior to screening or during the study without the prior written consent of the Medical Monitor.
6. Gastrointestinal, liver, kidney or other conditions which could interfere with the absorption, distribution, metabolism or excretion of Q-122 at PI discretion.
7. Untreated overt hyperthyroidism.
8. Have any other medical condition, clinically important systemic disease or significant co-morbidities or any finding during Screening that in the judgment of the investigator puts the participant at increased risk by participation in this study, or that may affect the reliability of participant diary entries.
9. Known inability to complete all study visits and study assessments for scheduling or other reasons.
10. BMI > 40 kg/m2; Participants with a BMI greater than 40 kg/m2 may be enrolled on a case-by-case basis if approved by the Medical Monitor and if the participant is not deemed at increased risk of adverse effects based on body habitus and cardiovascular health.
11. Women with a history of, or current evidence of, abuse of alcohol or any drug substance, or who regularly drink more than 3 standard drinks per day.
12. Uncontrolled systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥95 mmHg on 3 consecutive readings within the screening visit.
13. Abnormal laboratory findings:

    1. Hemoglobin < 9.5 g/dL (g/L); or any abnormal values that are deemed clinically significant by the investigator should be discussed with the medical monitor before being deemed ineligible.
    2. Fasting ALT, AST, GGT, or bilirubin greater than twice the upper limit of normal that is confirmed on a second sample.
    3. <60 eGFR mL/min/1.73 m2.
14. In the opinion of the investigator, have substantial risk of disease progression within the 3 months following screening and/or who potentially may require further treatment for their breast cancer during the study period including follow-up.
15. Any other reason which in the investigator's opinion makes the participant unsuitable for a clinical trial.
16. On any medications, either prescription or over-the-counter that are being taken solely for the purpose of treating VMS including SSRI/SNRI, gabapentin or pregabalin.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 132 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Hot Flash Severity Score (HFSS) | 4 weeks
  The primary efficacy outcome measure will be the change from baseline in the HFSS for moderate and severe hot flashes (HFSS-m/s) calculated for each treatment week by multiplying the severity by the frequency using the following formula: (2 x number of moderate) + (3 x number of severe)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (6):
  - North Georgia Clinical Research, Woodstock, Georgia
  - Indiana University School of Nursing, Indianapolis, Indiana
  - John Hopkins, Baltimore, Maryland
  - Brighams and Women's Hospital, Boston, Massachusetts
  - Stony Brook University, Stony Brook, New York
  - Baylor Scoot & White Medical Center, Temple, Texas
- Australia (7):
  - Royal Adelaide Hospital, Adelaide
  - ICON Group, Icon Cancer Care Wesley, Brisbane
  - School of Public Health and Preventive Medicine, Monash University, Melbourne
  - The Royal Women's Hospital, Melbourne
  - Keogh Institute for Medical Research, Perth
  - Women's Health Research Institute of Australia, Sydney
  - Royal North Shore Hospital, Sydney
- New Zealand (5):
  - Optimal Clinical Trials, Auckland
  - Auckland City Hospital, Auckland
  - Christchurch Clinical Studies Trust Ltd, Christchurch
  - P3 Research - Hawkes Bay, Havelock North
  - P3 Research - Tauranga, Tauranga

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vrselja A, Latifi A, Baber RJ, Stuckey BGA, Walker MG, Stearns V, Hickey M, Davis SR. Q-122 as a novel, non-hormonal, oral treatment for vasomotor symptoms in women taking tamoxifen or an aromatase inhibitor after breast cancer: a phase 2, randomised, double-blind, placebo-controlled trial. Lancet. 2022 Nov 12;400(10364):1704-1711. doi: 10.1016/S0140-6736(22)01977-8. PMID 36366886